CLINICAL TRIAL: NCT05655117
Title: Application of Artificial Intelligence in Early Detection of Eye Complications in Diabetics: A Randomized Clustered Trial in Hail, Saudi Arabia
Brief Title: Application of Artificial Intelligence in Early Detection of Eye Complications in Diabetics
Acronym: AI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The New Model of Care, Hail Health Cluster (Other Government)
Collaborators: Health Holding Company, Hail Health Cluster (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Model of Care Hail Cluster
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Artificial Intelegence; Diabetic Retinopathy Associated With Type 2 Diabetes Mellitus; Macular Edema Due to Type 2 Diabetes Mellitus
Keywords: AI Eye Screening in diabetics; Diabetic retinopathy; macular oedema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-based screening for early detection of diabetic retinopathy and macular Oedema (Experimental): The application of AI devices i.e Fundus Camera to detect diabetic retinopathy and macular Oedema in diabetics at the primary care centre
  Interventions: Other: AI based eye screening
- Routine screening for diabetic retinopathy and macular oedema (No Intervention): The Routine screening for diabetic retinopathy and macular oedema in diabetics during a routine visit to an eye care clinic at the primary care centre.

INTERVENTIONS:
Other: AI based eye screening — The application of AI devices i.e Fundus Camera to detect diabetic retinopathy and macular Oedema in diabetics at the primary care centre
  Arms: AI-based screening for early detection of diabetic retinopathy and macular Oedema

SUMMARY:
The goal of this pragmatic trial is to test the benefit of using artificial intelligence-based eye screening i.e, a fundus camera device in the early detection of eye complications in diabetics. The main questions it aims to answer are:

To what extent does the application of artificial intelligence-based eye care at primary care clinics work well in achieving early detection of eye complications such as macular oedema? To what extent does the application of artificial intelligence-based eye care at primary care clinics work well in achieving early detection of eye complications such as retinopathy? Participants will be asked to participate in the screening for eye complications at primary care centres, and a fundus camera will be used for screening.

Researchers will compare the proportion of detected cases with early signs of eye complication among those using artificial intelligence-based eye screening i.e., fundus camera, to the proportion of detected cases among those using routine eye care clinics at the primary care centre.

Early detection of eye complications in diabetics prevents the risk of blindness.

DETAILED DESCRIPTION:
In the era of artificial inelegance(AI), a shift from tertiary to secondary and primary care when caring for a patient with diabetic retinopathy is highly recommended.

Due to low operation, AI could be used in the early detection and screening of diabetic retinopathy by application of the service across a mass population and resource-limited areas with a scarcity of eye care services.

AI-based eye care in terms of screening for diabetic retinopathy will make the screening process more effective and cheap and could be delegated to technicians, practitioners, and/or even home-based self-screening.

Recognizing the high prevalence of type 2 diabetes mellitus (T2DM) among adults, the use of a nonmydriatic fundus camera with AI is effective in eye exams as it improves adult adherence to eye screening.

The primary aim of the trial will be to assess the effectiveness of the application of AI devices in terms of fundus cameras in the early detection of diabetic retinopathy and macular oedema among diabetic patients attending primary care centres.

Research Questions:

To what extent does the application of artificial intelligence-based eye care at primary care centre is effective in achieving a high detection rate of macular oedema? To what extent does the application of artificial intelligence-based eye care at primary care clinic is effective in achieving a high detection rate of retinopathy?

General objective:

To estimate the effectiveness of applying AI-based eye care at primary care centres in achieving a high detection rate of macular oedema and retinopathy among diabetics.

Specific Objectives:

Aim 1: To compare the proportion of detected cases of macular oedema in the intervention versus the control group (routine eye care) attending the primary care centre.

Aim 2: To compare the proportion of detected cases of retinopathy in the intervention versus the control group (routine eye care) attending the primary care centre

Literature Review:

Although recent models had been suggested for implementing digital health solutions like stream fishing, inflow funnel, pyramid, and shuffling cards that represent options for clinical services with progressively increasing capacity and willingness to operationalize digital health.

However, various challenges are facing the deployment of AI, telehealth, and the internet of things (IoT) worldwide. Barriers to adopting these digital health solutions are many and could be inferred to infrastructure, the quality of the device, common willingness, and legal aspects.

Evidence revealed that using Macustat retina function scan AI in remote monitoring of a patient with age-related macular oedema or diabetic retinopathy has a great impact on patient health.

Research Design and Methods:

This is a six months clustered randomized trial that will recruit patients with type II diabetes who are attending primary eye care clinics at primary care centres in Hail city.

Participants (P):

The participants will be type II diabetic patients of both genders attending the selected primary care centres irrespective of their duration of disease and the types of medication currently received. The participants are expected to be adults aged 18 years and above. Children and young adults with juvenile diabetes mellitus will be excluded. In addition, severely ill patients, and patients with mental disorders will be excluded. The participants will be assessed at the start to collect the baseline data about diabetic retinopathy and macular oedema using AI devices to report detected cases. At the end of the trial, a similar report of detected cases will be obtained three and six months after the beginning of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients aged 18-90

Exclusion Criteria:

* Severely ill patient or patient with cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The detection rate of diabetic retinopathy in the intervention group vs. control group | 6 month from the start of the study
  The proportion of the detected cases of diabetic retinopathy in the intervention group vs. control group
The detection rate of macular oedema in the intervention group vs. control group. | 6 month from the start of the study
  The proportion of the individuals who screened positive for macular oedema in the intervention group vs. control group.

SECONDARY OUTCOMES:
The screening rate for retinopathy | 6 months after the start of the study
  The proportion of individuals who receive eye care screening for diabetic retinopathy in the intervention group vs. control group.
The screening rate for macular odema | 6 months after the start of the study
  The proportion of individuals who receive eye care screening for macular oedema in the intervention group vs. control group

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Alshammari, VIP Chief MO, Study Chair — Hail Health Cluster; Fakhralddin Elfakki, Researcher at MOC, Principal Investigator — New Model of Care, Hail Health Cluser; Meshari Aljamani, MOC Lead, Study Director — New Model of Care, Hail Health Cluster

IPD SHARING:
Plan to Share IPD: No